CLINICAL TRIAL: NCT03495362
Title: The Effect of Insoluble Yeast Beta-glucan Intake on Pre-diabetic Patients: a Randomized Double-blind Trial
Brief Title: The Effect of Insoluble Yeast Beta-glucan Intake on Pre-diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHW20180201
Record Dates: First submitted 2018-03-22; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Pre-diabetic
Keywords: Yeast Beta-glucan; Immune Function; Prediabetes; Gut Microbiota
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The all details of groups assignment are arranged and controlled by the research designers. The color, shape, and external packaging of the yeast beta-glucan and placebo are consistent. Each bottle of capsules will be marked with the name (or identify number) of the participants by research designers. Thus, the grouping of participants is blind to the rest of the researchers (like outcomes assessors).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Ingredients: yeast beta-glucan, and capsule shell Capsule, per capsule with 500mg insoluble beta-glucan, twice a day, 1 capsule each time.
  The intervention period is about 3 months.
  Interventions: Dietary Supplement: Yeast Beta-glucan
- Placebo group (Placebo Comparator): Ingredients: starch, and capsule shell Capsule, per capsule with 500mg starch, twice a day, 1 capsule each time. The intervention period is about 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Yeast Beta-glucan — Twice a day, 1 capsule each time. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Intervention group
Other: Placebo — Twice a day, 1 capsule each time. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Placebo group

SUMMARY:
There is a lot of evidence to show that the yeast beta-glucan has immunomodulatory, anti-inflammatory, anti-infective effects.However,few work was done on the relationship between yeast bata-glucan and the immune function of diabetic patients. This is a randomized double-blind trial, aiming to study the effect of yeast beta-glucan on immune system of prediabetic patients. Firstly, the investigators will go into the efficacy of yeast beta-glucan on improving the clinical symptoms of prediabetics. Secondly, the investigators will study the mechanism of yeast beta-glucan on enhancing the immune function and improving the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years
* Meet the pre-diabetes diagnostic criteria recommended by World Health Organization (WHO) in 1999

Exclusion Criteria:

* Allergic to test substances
* Known severe heart, liver, kidney, autoimmune diseases, psychosis, nervous system, hematopoietic system, endocrine and other systemic diseases
* Known acute disease, common cold, metabolic diseases, chronic inflammation, infectious diseases, and heavy physical labor recently
* Usage of antihyperlipidemia or antihypertension, and other drugs may influence the interventional effect last two weeks
* Unable to cooperate with researchers or maintain ordinary dietary habit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Changes in the differentiation rates of some peripheral blood mononuclear cells (PBMCs) | At 0 week, 6th week, 12th week in the intervention period.
  Extract and isolate PBMCs from participants. Using flow cytometry to detect the differentiation rates of some PBMCs（Peripheral Blood Mononuclear Cells）inculding T, B, NK, CD4+, CD8+, CD19+, CD138+, CD3+ and CD45+ cells
Changes in inflammatory factors | At 0 week, 6th week, 12th week in the intervention period.
  Using ELISA to detect the expression level of TNF-α, IL-6, IL-1β, IL-12, IL-10, TGF-β
Changes in blood glucose level | At 0 week, 12th week in the intervention period.
  FPG(fasten plasma glucose), OGTT（oral glucose tolerance test）
Changes in gut microbiota | At 0 week, 6th week, 12th week in the intervention period.
  High-throughput 16S DNA gene amplicon sequencing performed on the Illumina HiSeq platform.
Changes in RTI(respiratory tract infection) | Every week across the intervention peroid，an average of 3 months.
  Observe the clinical symptoms of respiratory infections in two groups of patients
Changes in islet function | At 0 week, 12th week in the intervention period.
  C-peptide level

SECONDARY OUTCOMES:
Changes in SCFA (short chain fatty acids) | At 0 week, 6th week, 12th week in the intervention period.
  Using GC-MS to detect fecal and plasma SCFA
Changes in blood lipids profile | At 0 week, 12th week in the intervention period.
  Fasting plasma Total cholesterol, Low Density Lipoprotein, High Density Lipoprotein and triglycerides.
Changes in hepatorenal function | At 0 week, 12th week in the intervention period.
  Using automatic biochemical analyzer to detect creatinine, urea nitrogen, alanine aminotransferase, aspartate aminotransferase and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided